CLINICAL TRIAL: NCT03808909
Title: Providing Expanded Continuous Labor Support to Pregnant Women in New Mexico With Substance Use Disorders
Acronym: Project_SuM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Pilar Sanjuan, Research Assistant Professor, University of New Mexico
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 18-280; 5U54MD004811-10 (NIH)
Record Dates: First submitted 2019-01-14; First posted 2019-01-18 (Actual); Results first posted 2022-11-30 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Pregnancy Related; Substance Use Disorders
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Doula (Experimental): Participants will be assigned a doula.
  Interventions: Other: Continuous Labor Support
- Control (No Intervention): Participants will not be assigned a doula.

INTERVENTIONS:
Other: Continuous Labor Support — Participants in the intervention condition will be assigned a doula who is a lay person trained to provide emotional and practical support to individuals throughout labor and delivery.
  Arms: Doula

SUMMARY:
This study will determine the feasibility of offering expanded continuous labor support by trauma- and addiction-trained medical paraprofessionals (i.e. doulas) at no cost to pregnant women receiving care for substance use disorders (SUD). The long-term goal of this transdisciplinary multilevel intervention is ultimately to reduce a major existing behavioral health disparity in the state. This cross-campus multi-disciplinary collaboration, is in partnership with Young Women United (a research and policy organization in NM) and doulas of the UNM Birth Companion Program. Through this partnership, women receiving combined OB/SUD treatment at the Milagro Program at UNMHSC will be offered expanded doula services.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years old
* able to participate in informed consent
* able to read, write, and speak English
* gestation of at least 26 weeks at baseline (necessary because of short duration of study)
* plan to give birth at UNM.

Exclusion Criteria:

* active psychosis
* current incarceration
* identified by medical staff as unable for medical reasons to currently participate in the study
* not interested in having doula support

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2019-02-06 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-07-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of New Mexico, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Doula | Control
Started | 12 | 1
Completed | 9 | 1
Not Completed | 3 | 0
Not completed — Lost to Follow-up | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Doula | Control | Total
Number analyzed (Participants) | 9 | 1 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 1 | 10
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 1 | 10
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 1 | 7
  Not Hispanic or Latino | 3 | 0 | 3
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 8 | 1 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 9 | 1 | 10
Edinburgh Postpartum Depression Scale [Mean (Standard Deviation); unit: units on a scale] | 12.11 (5.6667) | 18 (0) | 12.70 (5.65784)
PTSD Checklist - 5 (PCL-5) [Mean (Standard Deviation); unit: units on a scale] — The PCL-5 is a 20-item questionnaire, corresponding to the DSM-5 symptom criteria for PTSD. The wording of PCL-5 items reflects both changes to existing symptoms and the addition of new symptoms in DSM-5.
  A total symptom severity score (range - 0-80) can be obtained by summing the scores for each of the 20 items.
  Initial research suggests that a PCL-5 cutoff score between 31-33 is indicative of probable PTSD across samples.
  See: https://www.ptsd.va.gov/professional/assessment/adult-sr/ptsd-checklist.asp
  units on a scale | 35.56 (23.591) | 23 (0) | 34.30 (22.593)
Percent Drinking Days [Mean (Standard Deviation); unit: Percent of days] — Percent drinking days from pregnancy recognition to baseline assessment collected with the Timeline Followback. See SOBELL, L.C., SOBELL, M.B., LEO, G.I. and CANCILLA, A. (1988), Reliability of a Timeline Method: assessing normal drinkers' reports of recent drinking and a comparative evaluation across several populations. British Journal of Addiction, 83: 393-402. https://doi-org.libproxy.unm.edu/10.1111/j.1360-0443.1988.tb00485.x
  Percent of days | 0 (0) | 0 (0) | 0 (0)
Percent Substance Use Days [Mean (Standard Deviation); unit: Percent of days] — Sum of all percent substance use days - can be more than 100% if multiple substances used during the same time frame (from pregnancy recognition to baseline assessment). SOBELL, L.C., SOBELL, M.B., LEO, G.I. and CANCILLA, A. (1988), Reliability of a Timeline Method: assessing normal drinkers' reports of recent drinking and a comparative evaluation across several populations. British Journal of Addiction, 83: 393-402. https://doi-org.libproxy.unm.edu/10.1111/j.1360-0443.1988.tb00485.x
  Percent of days | 52.75 (56.372) | 0 (0) | 47.47 (55.704)
NIH Toolbox Emotional Support [Mean (Standard Deviation); unit: units on a scale] — Measures perceived emotional support. Scale range = 5-40. Higher scores indicate more perceived support. See https://www.healthmeasures.net/explore-measurement-systems/nih-toolbox
  units on a scale | 33.00 (6.727) | 9 (0) | 30.60 (9.891)
NIH Toolbox Friendship Support [Mean (Standard Deviation); unit: units on a scale] — Measures perceived support from friends. Scale range = 5-40. Higher scores indicate more perceived support from friends. See: https://www.healthmeasures.net/explore-measurement-systems/nih-toolbox
  units on a scale | 17.89 (5.578) | 8 (0) | 16.90 (6.118)
NIH Toolbox Instrumental Support [Mean (Standard Deviation); unit: units on a scale] — Measures perceived instrumental support. Range = 5-40. Higher scores indicate more perceived support. See https://www.healthmeasures.net/explore-measurement-systems/nih-toolbox
  units on a scale | 29.22 (5.740) | 8 (0) | 27.10 (8.621)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Remain in the Study
Description: Number of participants who complete the 2 week follow-up
Time Frame: 2 week postpartum follow-up assessment
Measure: Count of Participants; unit: Participants
Arm/Group | Doula | Control
Number analyzed (Participants) | 9 | 1
Participants | 9 | 1

2. Secondary Outcome: Alternative Birth Outcome
Description: Number of participants with preterm, c-section, fetal demise, still birth, or other potential birth outcomes
Time Frame: birth
Measure: Count of Participants; unit: Participants
Arm/Group | Doula | Control
Number analyzed (Participants) | 9 | 1
Participants
  C-section | 2 | 1
  Preterm Birth | 1 | 0
  Fetal Demise | 0 | 0
  Stillbirth | 0 | 0

3. Secondary Outcome: Postpartum Posttraumatic Stress Disorder Checklist
Description: PTSD Checklist - 5 (PCL-5) Higher scores indicate a worse outcome Range of scale = 0 - 80
Time Frame: 2 week postpartum follow-up assessment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Doula | Control
Number analyzed (Participants) | 9 | 1
score on a scale | 21.38 (20.007) | 50 (0)

4. Secondary Outcome: Participant Satisfaction
Description: Study specific participant satisfaction - debriefing form - qualitative data. No qualitative analyses have been conducted with this data.
Time Frame: 2 week postpartum follow-up assessment
Population: Participants who were assigned a doula were included in this analysis
Measure: Number; unit: percentage of participants
Arm/Group | Doula | Control
Number analyzed (Participants) | 9 | 0
percentage of participants
  Percent of participants who found it very helpful emotionally to have a doula during labor/delivery | 89 |
  Percent of participants who found it very helpful physically to have a doula during labor/delivery | 89 |
  Percent of participants who found it very helpful socially to have a doula during labor/delivery | 100 |
  Percent of participants who would want a doula at another birth | 100 |
  Percent of participants who felt having a doula made pregnancy much easier | 89 |
  Percent of participants who felt the doula understood their needs very well | 89 |
  Percent of participants who were very satisfied with the doula experience | 100 |

5. Other Pre Specified Outcome: Percentage of Days With Drinking or Substance Use
Description: Using the timeline followback we will calculate average percentage of days of alcohol or other substance use for each group from pregnancy recognition to the 2 week follow-up.
Time Frame: 2 week postpartum follow-up assessment
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | Doula | Control
Number analyzed (Participants) | 9 | 1
percentage of days | 19.85 (44.509) | 0 (0)

6. Other Pre Specified Outcome: Mother's Autonomy During Birth
Description: Mother's Autonomy in Decision Making Questionnaire Higher scores indicate more autonomy (better outcome) Scale range = 7 - 42
Time Frame: queries feelings during labor and birth but is administered at 2 week follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Doula | Control
Number analyzed (Participants) | 9 | 1
score on a scale | 30.8889 (11.66667) | 38 (0)

7. Other Pre Specified Outcome: Postpartum Depression
Description: Edinburgh Postpartum Depression Scale Higher scores are a worse outcome Scale range = 0-30
Time Frame: 2 week postpartum follow-up assessment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Doula | Control
Number analyzed (Participants) | 9 | 1
score on a scale | 8.56 (6.579) | 18 (0)

8. Other Pre Specified Outcome: Breastfeeding Update
Description: Using a study specific form we will calculate the number of participants who attempted breastfeeding after the birth of the baby
Time Frame: 2 week postpartum follow-up assessment
Measure: Count of Participants; unit: Participants
Arm/Group | Doula | Control
Number analyzed (Participants) | 9 | 1
Participants
  Breastfeeding intent | 3 | 1
  Breastfeeding initiation | 9 | 1
  Breastfeeding at discharge | 9 | 1
  Exclusive breastfeeding | 2 | 0

9. Other Pre Specified Outcome: Neonatal Abstinence Syndrome
Description: NAS diagnosis
Time Frame: neonatal
Measure: Count of Participants; unit: Participants
Arm/Group | Doula | Control
Number analyzed (Participants) | 9 | 1
Participants | 6 | 0

10. Other Pre Specified Outcome: Length of NICU Stay
Description: Average length of time that the infant remains hospitalized in the NICU after the birth
Time Frame: from birth through study completion, an average of 3 months
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Doula | Control
Number analyzed (Participants) | 9 | 1
Days | 11.56 (14.32) | 4 (0)

11. Other Pre Specified Outcome: Social Support - NIH Toolbox
Description: Average score for social support on NIH toolbox Total of Emotional, Friend, and Instrumental Social support scales Higher scores indicated a better outcome Scale range = 24 - 120
Time Frame: 2 week postpartum follow-up assessment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Doula | Control
Number analyzed (Participants) | 9 | 1
score on a scale | 82.3333 (19.62142) | 25 (0)

ADVERSE EVENTS:
Description: Adverse event data was not collected as there was no data monitoring plan because this research was not considered more than minimal risk.
Groups:
- Doula: Participants with a doula
- No Doula: Participants without a doula
Arm/Group | Doula | No Doula
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
This was a pilot feasibility study. We only collected data for 10 participants: 9 in the experimental condition - with a doula and 1 in the control condition. Thus, the data is primarily descriptive and there are not enough participants to conduct statistical comparisons between groups. This was because funding was only available for 12 mos and negotiations between community partners and the university delayed the start of data collection by more than 6 months.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-12): https://cdn.clinicaltrials.gov/large-docs/09/NCT03808909/Prot_SAP_000.pdf